CLINICAL TRIAL: NCT04745520
Title: Comparison of Rib Fixation with Medical Analgesia in Patients with Uncomplicated Rib Fractures on Pain Control: a Multi-center Randomized Clinical Trial
Brief Title: Randomized Clinical Trial of Rib Fixation Versus Medical Analgesia in Uncomplicated Rib Fractures on Pain Control.
Acronym: PAROS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Participant recruitment was too low. One of the reasons is the overly strict exclusion criteria.
Sponsor: Benoît Bédat (Other)
Collaborators: Centre Hospitalier Universitaire Vaudois (Other); Hôpital du Valais (Other)
Responsible Party: Sponsor-Investigator, Benoît Bédat, Fellow, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-01688
Record Dates: First submitted 2020-12-06; First posted 2021-02-09 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Rib Fractures
Keywords: thoracic trauma; rib fixation; medical device
MeSH Terms: conditions — Rib Fractures | interventions — Analgesia

STUDY DESIGN:
Intervention Model Description: This pragmatic trial is a multi-center, two-arm, parallel-group, superiority randomized-controlled trial.
Masking Description: it is not possible to blind the patients and investigators regarding surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rib fixation (medical devices) (Experimental): Surgery and pain medication. The pain of patients will be treated with rib fixation and pain medication.
  Interventions: Device: Rib fixation; Drug: Analgesia
- Pain medication (comparator treatment) (Active Comparator): Pain medication only.
  Interventions: Drug: Analgesia

INTERVENTIONS:
Device: Rib fixation — Rib fixation is performed by a senior surgeon. The patient is under general anesthesia. A thoracotomy focused on the fracture is performed to optimize access to the rib to be repaired. Video-assisted thoracic surgery (VATS) can be performed to better localize rib fractures. Significant muscle division is avoided. Removal of the periosteum is not required. The broken rib segments are approximated with forceps and the medical devices are used to fix the fracture. The medical devices are implemented according to the manufacturers' recommendations. The goal is to stabilize the chest wall. It is not useful to fix all fractures to stabilize the wall. A chest tube can be placed at the end of the operation.
  Medical devices
  The following medical devices can be used:
  * MatrixRIB™, De Puy Synthes Companies, Zuchwill, Switzerland
  * STRATOS™, MedXpert GmbH, Heitersheim, Germany
  * NiTi Fixing PlatesTM, IAWAI, Yandzhou, China
  Arms: Rib fixation (medical devices)
Drug: Analgesia — Epidural analgesia is continuing for 24 to 72 hours post-randomization to maximize outcome benefits. Afterwards, paracetamol, NSAID and/or opioid treatment are used according to pain severity. In case of opioid use, morphine treatment is preferred. However, other opioid drugs or doses can be considered to better customize the treatment.

SUMMARY:
Uncomplicated costal fractures often result in persistent pain over the long term. Indeed, cohort studies showed that at 6 months, 22% of patients still had pain and 56% had functional disability. The impact of costal fractures on quality of life is underestimated. The socio-psycho-economic consequences are substantial.

Previous studies have shown that an important factor for persistent pain and functional disability is the intensity of the initial pain. However, preliminary studies have shown promising results with surgical fixation of rib fractures: reduced need for analgesic drugs, reduced pain at 1 month, reduced complications and improved motor skills in patients over 65 years of age.

To date, the only clinical trials that exist focused on the fixation of complicated rib dislocations. While fixation of uncomplicated rib fractures is a common practice, no randomized studies have been conducted to evaluate its impact on pain and quality of life in the medium and long term.

In this context, the aim of our randomized study is to compare pain at 2 months between operated and non-operated patients with uncomplicated rib fractures.

DETAILED DESCRIPTION:
Background. Until recently, functional disability and chronic pain and following uncomplicated rib fractures have been scarcely studied. Studies described persistent pain and disability in, respectively, 59% and 76% of patients at two months, and in 22% and 53% of patients at 6 months. In a retrospective study including 216 patients with an isolated thoracic injury, only 34.2% of patients had a good recovery at one year and the six-month return to work rate is of 63%. Persistent pain and disability following rib fractures therefore result in a large psycho-socio-economic impact for health-care system. The only predictive factor for persistent pain and disability is the pain intensity within the first few days after injury. Similarly, the intensity of pain within the first days after thoracotomy predicts long-term post-thoracotomy pain. In a recent meta-analysis, epidural analgesia provides better acute pain relief than intravenous, paravertebral, and intercostal interventions. While meta-analyses conclude that operative fixation of complicated flail chest provide better outcome, the impact of surgery on pain in uncomplicated rib fracture is seldom studied. Some retrospective studies showed promising results of rib fixation with surgery in patients with uncomplicated rib fractures: A study showed that rib fixation reduced postoperative analgesic requirements. Similarly, another study showed that pain was significantly reduced one month after surgery as compared to a non-surgical approach. Finally, it has been recently observed a decreased mortality and respiratory complications after surgery in patients over 65 years old as well as a better functional status at two weeks, two months, and four months.

Trial objectives. No previous studies have provided definitive evidence for recommending rib fixation over simple pain medication to control pain. Our hypothesis is that a surgical approach may have further benefits as compared to a conservative treatment. The primary objective of the study is to compare pain two months after injury between two groups: group 1) patients who are treated with surgery and analgesic treatment; and group 2) patients who are treated with analgesic treatment alone. The secondary objective is to perform a longitudinal analysis over one year of the following parameters: amount of pain medication, quality of life, anxiety and depression, pulmonary capacity, return to work, and adverse events. Financial aspects are also investigated.

ELIGIBILITY:
Inclusion Criteria:

* At least 2 rib fractures
* At least 1 dislocated rib fracture
* Fractures accessible to surgery
* Thoracic trauma no more than two days prior to screening for inclusion
* Thoracic epidural analgesia
* Written informed consent

Exclusion Criteria:

* Any other concomitant fractures excepted clavicle fracture
* Respiratory distress syndrome according to the Berlin definition
* Presence of >1.5 liter of blood drained from the pleural space
* Hemostasis disorder defined by any of the following criteria:

  * Platelet count < 70'000/mm3,
  * International Normalized Ratio (INR) > 1.2 (Prothrombin < 70%)
  * activated partial thromboplastin time (aPTT) ≥ 60 seconds
  * drugs such as: P2Y12 antagonists (clopidogrel, prasugrel) and glycoprotein IIb/IIIa antagonists (abciximab, tirofiban)
* Pathological rib fracture due to metastasis
* Hemodynamic instability: systolic blood pressure < 100 mmHg and heart rate > 100 beats per minute
* Neurologic disorder: Glasgow Coma Score < 13 in the initial 24 hours, or intracerebral, epidural, subdural, or subarachnoid hemorrhages, or cerebral contusion
* Titanium allergy
* Known or suspected non-compliance to medical therapy due to drug or alcohol abuse
* Age <18 years old
* Women who know they are pregnant or breast feeding
* Inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2021-03-12 (Actual); Primary Completion 2023-11-16 (Actual); Study Completion 2024-09-16 (Actual)

PRIMARY OUTCOMES:
Pain severity | Two months after injury
  Pain level reported by the participant, as assessed via the first part of the French version of the brief pain inventory (BPI) questionnaire. 0-10 scale. 10 indicating worst pain

SECONDARY OUTCOMES:
Pain severity | At recruitment (baseline)
  Pain level reported by the participant, as assessed via the first part of the French version of the brief pain inventory (BPI) questionnaire. 0-10 scale. 10 indicating worst pain
Pain severity | One month after injury
  Pain level reported by the participant, as assessed via the first part of the French version of the brief pain inventory (BPI) questionnaire. 0-10 scale. 10 indicating worst pain
Pain severity | Three months after injury
  Pain level reported by the participant, as assessed via the first part of the French version of the brief pain inventory (BPI) questionnaire. 0-10 scale. 10 indicating worst pain
Pain severity | Six months after injury
  Pain level reported by the participant, as assessed via the first part of the French version of the brief pain inventory (BPI) questionnaire. 0-10 scale. 10 indicating worst pain
Pain severity | Twelve months after injury
  Pain level reported by the participant, as assessed via the first part of the French version of the brief pain inventory (BPI) questionnaire. 0-10 scale. 10 indicating worst pain
Anxiety and Depression. | At recruitment (baseline)
  hospital anxiety and depression scale (HADS). Score 0-21. 21 = severe depression or anxiety
Anxiety and Depression. | One month after injury
  hospital anxiety and depression scale (HADS). Score 0-21. 21 = severe depression or anxiety
Anxiety and Depression. | Two months after injury
  hospital anxiety and depression scale (HADS). Score 0-21. 21 = severe depression or anxiety
Neuropathic pain | Two months after injury
  The French questionnaire "Douleur Neuropathique en 4 Questions (DN4)" is completed by an investigator during follow-up visits. The DN4 questionnaire was developed to diagnose polyneuropathy. Three items are linked with neuropathic pain examination, and seven items to pain symptoms. Score 0-10. Score >4 indicates neuropathic pain.
Neuropathic pain | Six months after injury
  The French questionnaire "Douleur Neuropathique en 4 Questions (DN4)" is completed by an investigator during follow-up visits. The DN4 questionnaire was developed to diagnose polyneuropathy. Three items are linked with neuropathic pain examination, and seven items to pain symptoms. Score 0-10. Score >4 indicates neuropathic pain.
Pain interference | At recruitment (baseline)
  The last items of the BPI questionnaires measure how much pain has interfered with seven daily activities, including general activity, walking, work, mood, enjoyment of life, relations with others and sleep. BPI pain interference is scored as the mean of the seven items. Score 0-10. 10 = high interference of pain with activities.
Pain interference | One month after injury
  The last items of the BPI questionnaires measure how much pain has interfered with seven daily activities, including general activity, walking, work, mood, enjoyment of life, relations with others and sleep. BPI pain interference is scored as the mean of the seven items. Score 0-10. 10 = high interference of pain with activities.
Pain interference | Two months after injury
  The last items of the BPI questionnaires measure how much pain has interfered with seven daily activities, including general activity, walking, work, mood, enjoyment of life, relations with others and sleep. BPI pain interference is scored as the mean of the seven items. Score 0-10. 10 = high interference of pain with activities.
Pain interference | Three months after injury
  The last items of the BPI questionnaires measure how much pain has interfered with seven daily activities, including general activity, walking, work, mood, enjoyment of life, relations with others and sleep. BPI pain interference is scored as the mean of the seven items. Score 0-10. 10 = high interference of pain with activities.
Pain interference | Six months after injury
  The last items of the BPI questionnaires measure how much pain has interfered with seven daily activities, including general activity, walking, work, mood, enjoyment of life, relations with others and sleep. BPI pain interference is scored as the mean of the seven items. Score 0-10. 10 = high interference of pain with activities.
Pain interference | Twelve months after injury
  The last items of the BPI questionnaires measure how much pain has interfered with seven daily activities, including general activity, walking, work, mood, enjoyment of life, relations with others and sleep. BPI pain interference is scored as the mean of the seven items. Score 0-10. 10 = high interference of pain with activities.
Health and well being | At recruitment (baseline)
  The 36-Item Health Survey (SF-36) taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. Score: 0-100. 100 = better functioning
Health and well being | Two months after injury
  The 36-Item Health Survey (SF-36) taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. Score: 0-100. 100 = better functioning
Health and well being | Six months after injury
  The 36-Item Health Survey (SF-36) taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. Score: 0-100. 100 = better functioning
Analgesic medication during hospitalisation | At recruitement (baseline)
  During hospitalization, each day since the enrolment, amount and type of analgesic medication are recorded from the computerized patient record system.
Analgesic medication at home | One month after injury
  After discharge, analgesic medication (type and amount) is tracked using a custom questionnaire.
Analgesic medication at home | Two months after injury
  After discharge, analgesic medication (type and amount) is tracked using a custom questionnaire.
Analgesic medication at home | Three months after injury
  After discharge, analgesic medication (type and amount) is tracked using a custom questionnaire.
Analgesic medication at home | Six months after injury
  After discharge, analgesic medication (type and amount) is tracked using a custom questionnaire.
Analgesic medication at home | Twelve months after injury
  After discharge, analgesic medication (type and amount) is tracked using a custom questionnaire.
Productivity & return to work | One month after injury
  The work productivity and activity impairment (WPAI) questionnaire is used. It assesses impairments in both paid work and unpaid work. It measures absenteeism, presenteeism as well as the impairments in unpaid activity because of health problem during the past seven days. Score 0-10. 10 = high impairment
Productivity & return to work | Two months after injury
  The work productivity and activity impairment (WPAI) questionnaire is used. It assesses impairments in both paid work and unpaid work. It measures absenteeism, presenteeism as well as the impairments in unpaid activity because of health problem during the past seven days. Score 0-10. 10 = high impairment
Productivity & return to work | Three months after injury
  The work productivity and activity impairment (WPAI) questionnaire is used. It assesses impairments in both paid work and unpaid work. It measures absenteeism, presenteeism as well as the impairments in unpaid activity because of health problem during the past seven days. Score 0-10. 10 = high impairment
Productivity & return to work | Six months after injury
  The work productivity and activity impairment (WPAI) questionnaire is used. It assesses impairments in both paid work and unpaid work. It measures absenteeism, presenteeism as well as the impairments in unpaid activity because of health problem during the past seven days. Score 0-10. 10 = high impairment
Productivity & return to work | Twelve months after injury
  The work productivity and activity impairment (WPAI) questionnaire is used. It assesses impairments in both paid work and unpaid work. It measures absenteeism, presenteeism as well as the impairments in unpaid activity because of health problem during the past seven days. Score 0-10. 10 = high impairment
Pulmonary function | Two months after injury
  Forced vital capacity (FVC, % predicted) measured according to the recommendations of the European Respiratory Society. The best value of at least three tests is recorded.
Pulmonary function, forced vital capacity | Six months after injury
  Forced vital capacity (FVC, % predicted) measured according to the recommendations of the European Respiratory Society. The best value of at least three tests is recorded.
Pulmonary function, peak expiratory flow | Two months after injury
  Peak expiratory flow (PEF, L/min) measured according to the recommendations of the European Respiratory Society. The best value of at least three tests is recorded.
Pulmonary function, peak expiratory flow | Six months after injury
  Peak expiratory flow (PEF, L/min) measured according to the recommendations of the European Respiratory Society. The best value of at least three tests is recorded.
Pulmonary function, sniff nasal inspiratory pressure | Two months after injury
  sniff nasal inspiratory pressure (in in cmH2O) measured according to the recommendations of the European Respiratory Society. The best value of at least three tests is recorded.
Pulmonary function, sniff nasal inspiratory pressure | Six months after injury
  sniff nasal inspiratory pressure (in in cmH2O) measured according to the recommendations of the European Respiratory Society. The best value of at least three tests is recorded.
Pulmonary function, inspiratory pressure | Two months after injury
  Maximum inspiratory pressure (in in cmH2O) measured according to the recommendations of the European Respiratory Society. The best value of at least three tests is recorded.
Pulmonary function, inspiratory pressure | Six months after injury
  Maximum inspiratory pressure (in in cmH2O) measured according to the recommendations of the European Respiratory Society. The best value of at least three tests is recorded.
Length of hospital stay | from admission to discharge, up to four weeks
  Length of hospital stay is reported in days from the day of hospitalization until the hospital discharge. The length of convalescence stay is also reported.
Total costs | Twelve months after injury
  Costs are reported at the end of the follow-up period (12 months) in swiss francs. They include costs for hospital treatment and costs for medication.
Adverse events | From inclusion to the end of the study, up to 12 months
  We collect safety outcomes in accordance with international standards (ISO 14155 and ICH-GCP)

CONTACTS AND LOCATIONS:
Overall Officials: Benoît Bédat, MD, Principal Investigator — University Hospital, Geneva; Frédéric Triponez, Prof., Study Chair — University Hospital, Geneva
Locations (1):
- Unit of Thoracic and Endocrine Surgery, University Hospitals of Geneva, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kerr-Valentic MA, Arthur M, Mullins RJ, Pearson TE, Mayberry JC. Rib fracture pain and disability: can we do better? J Trauma. 2003 Jun;54(6):1058-63; discussion 1063-4. doi: 10.1097/01.TA.0000060262.76267.EF. PMID 12813323
- [Background] Fabricant L, Ham B, Mullins R, Mayberry J. Prolonged pain and disability are common after rib fractures. Am J Surg. 2013 May;205(5):511-5; discusssion 515-6. doi: 10.1016/j.amjsurg.2012.12.007. PMID 23592156
- [Background] Gordy S, Fabricant L, Ham B, Mullins R, Mayberry J. The contribution of rib fractures to chronic pain and disability. Am J Surg. 2014 May;207(5):659-62; discussion 662-3. doi: 10.1016/j.amjsurg.2013.12.012. Epub 2014 Jan 31. PMID 24612969
- [Background] Marasco S, Lee G, Summerhayes R, Fitzgerald M, Bailey M. Quality of life after major trauma with multiple rib fractures. Injury. 2015 Jan;46(1):61-5. doi: 10.1016/j.injury.2014.06.014. Epub 2014 Jun 21. PMID 25069400
- [Background] Katz J, Jackson M, Kavanagh BP, Sandler AN. Acute pain after thoracic surgery predicts long-term post-thoracotomy pain. Clin J Pain. 1996 Mar;12(1):50-5. doi: 10.1097/00002508-199603000-00009. PMID 8722735
- [Background] de Moya M, Bramos T, Agarwal S, Fikry K, Janjua S, King DR, Alam HB, Velmahos GC, Burke P, Tobler W. Pain as an indication for rib fixation: a bi-institutional pilot study. J Trauma. 2011 Dec;71(6):1750-4. doi: 10.1097/TA.0b013e31823c85e9. PMID 22182884
- [Background] Wu WM, Yang Y, Gao ZL, Zhao TC, He WW. Which is better to multiple rib fractures, surgical treatment or conservative treatment? Int J Clin Exp Med. 2015 May 15;8(5):7930-6. eCollection 2015. PMID 26221350
- [Background] Fitzgerald MT, Ashley DW, Abukhdeir H, Christie DB 3rd. Rib fracture fixation in the 65 years and older population: A paradigm shift in management strategy at a Level I trauma center. J Trauma Acute Care Surg. 2017 Mar;82(3):524-527. doi: 10.1097/TA.0000000000001330. PMID 28030506
- [Background] Peek J, Smeeing DPJ, Hietbrink F, Houwert RM, Marsman M, de Jong MB. Comparison of analgesic interventions for traumatic rib fractures: a systematic review and meta-analysis. Eur J Trauma Emerg Surg. 2019 Aug;45(4):597-622. doi: 10.1007/s00068-018-0918-7. Epub 2018 Feb 6. PMID 29411048
- [Derived] Perentes JY, Christodoulou M, Abdelnour-Berchtold E, Karenovics W, Gayet-Ageron A, Gonzalez M, Krueger T, Triponez F, Terrier P, Bedat B. Effectiveness of rib fixation compared to pain medication alone on pain control in patients with uncomplicated rib fractures: study protocol of a pragmatic multicenter randomized controlled trial-the PAROS study (Pain After Rib OSteosynthesis). Trials. 2022 Sep 2;23(1):732. doi: 10.1186/s13063-022-06509-0. PMID 36056421